CLINICAL TRIAL: NCT02292004
Title: Bridge-Enhanced ACL Repair-Safety Study
Brief Title: Bridge-Enhanced ACL Repair-Safety Study (BEAR Trial)
Acronym: BEAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miach Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: IRB-P00012985
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Injury; Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ACL repair with MIACH scaffold (Experimental): Patients will undergo ACL repair surgery using the newly developed MIACH scaffold
  Interventions: Device: ACL Repair with MIACH Scaffold
- Standard ACL reconstruction (Active Comparator): Patients will undergo a standard ACL reconstruction surgery
  Interventions: Procedure: Standard ACL Reconstruction

INTERVENTIONS:
Device: ACL Repair with MIACH Scaffold — Surgical insertion of the MIACH scaffold to promote ACL healing/repair
  Arms: ACL repair with MIACH scaffold
Procedure: Standard ACL Reconstruction — Standard surgical reconstruction of the ACL with autograft hamstring tendon
  Arms: Standard ACL reconstruction

SUMMARY:
This study will assess the safety and early efficacy of a newly developed device, bridge-enhanced scaffold (MIACH™,) used to repair a torn anterior cruciate ligament (ACL.) Ten participants will undergo surgery with the new device (Experimental Group) and 10 will undergo a standard ACL reconstruction surgery (Control Group.)

DETAILED DESCRIPTION:
This is a first-in-human trial for evaluation of the safety (Primary Objective) and short-term efficacy (Secondary Objective) of the MIACH™ ACL scaffold and will be carried out in form of an observational study of 20 patients: 10 experimental and 10 control.

ELIGIBILITY:
Inclusion Criteria:

* Complete ACL tear, confirmed by MRI
* Time from injury to screening must be less than or equal to 90 days
* ACL tissue present on pre-operative MRI

Exclusion Criteria (before surgery):

* Prior surgery on affected knee
* History of prior infection in affected knee
* Regular use of tobacco or nicotine in any form
* Use of corticosteroid within last 6 months
* Ever underwent chemotherapy treatment
* History of sickle cell disease
* History of anaphylaxis
* Any condition that could affect healing (Diabetes, inflammatory arthritis, etc)
* Diagnosis of posterolateral corner injury (LCL complete tear, Biceps femoris tendon avulsion, tear of the arcuate ligament, tear of the popliteus ligament)
* Diagnosis of Grade III medial collateral ligament injury
* Diagnosis of complete patellar dislocation

Exclusion Criteria (during surgery):

* ACL deemed normal on arthroscopic inspection
* Time from injury to surgery is greater than 90 days (for Comparator group) and greater than 30 days (for Experimental group)
* Experimental Group: Less than 50 percent of ACL remaining
* Displaced bucket handle meniscal injury requiring repair
* Diagnosis of full-thickness chondral injury on either condyle
* Grade III medial collateral ligament injury

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of the BEAR® Implant | Surgery to 3-months post-op
  To assess the safety (implant rejection, infection, joint effusion, muscle atrophy, knee laxity) and tolerability of the BEAR® implant

SECONDARY OUTCOMES:
Inflammatory reaction | Surgery to 3-months post-op
  Tense effusion limiting motion, fever or increased knee pain for more than three weeks after surgery and synovial fluid culture is negative for organisms.
Muscle Atrophy | At 6-weeks post-op
  Patient cannot ambulate independently and continues to require crutches for ambulation for more than six weeks after surgery as a result of the muscle weakness. Patient report leg feels unstable ambulating without crutches at six weeks after surgery.
Excessive Pain | Surgery to 3-months post-op
  Patient needs to be readmitted to the hospital for parenteral (IV or IM) pain medications but no other adverse event (e.g. infection or inflammation) is found.
Implant failure | At 3-months post-op
  Lachman exam demonstrates 6mm or greater AP knee laxity when the knee is in 25 degrees of flexion in the operated knee than the unoperated knee on examination by the physician in the office. Both knees will be covered and the examining physician blinded to which knee was the surgical knee prior to the testing.
Anteroposterior (AP) knee laxity | At 6- and 12-months post-op
  KT-1000 testing of AP laxity in both knees reveals a side-to-side difference of >=6mm when performed by the clinician. The knees will be covered and the examiner blinded as to which is the operated knee.

CONTACTS AND LOCATIONS:
Overall Officials: Lyle Micheli, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall TL, Thompson RW. Interhemispheric transfer as a function of light intensity discrimination difficulty. J Comp Physiol Psychol. 1971 Oct;77(1):166-70. doi: 10.1037/h0031569. No abstract available. PMID 5120682
- [Derived] Barnett SC, Murray MM, Flannery SW; BEAR Trial Team; Menghini D, Fleming BC, Kiapour AM, Proffen B, Sant N, Portilla G, Sanborn R, Freiberger C, Henderson R, Ecklund K, Yen YM, Kramer D, Micheli L. ACL Size, but Not Signal Intensity, Is Influenced by Sex, Body Size, and Knee Anatomy. Orthop J Sports Med. 2021 Dec 17;9(12):23259671211063836. doi: 10.1177/23259671211063836. eCollection 2021 Dec. PMID 34988237
- [Derived] Kiapour AM, Ecklund K, Murray MM; BEAR Trial Team; Flutie B, Freiberger C, Henderson R, Kramer D, Micheli L, Thurber L, Yen YM, Fleming BC. Changes in Cross-sectional Area and Signal Intensity of Healing Anterior Cruciate Ligaments and Grafts in the First 2 Years After Surgery. Am J Sports Med. 2019 Jul;47(8):1831-1843. doi: 10.1177/0363546519850572. Epub 2019 Jun 5. PMID 31166701